CLINICAL TRIAL: NCT04433845
Title: The Safety and Efficacy of Psilocybin in Participants With Type 2 Bipolar Disorder (BP-II) Depression.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: COMPASS Pathways (Industry)
Responsible Party: Principal Investigator, Scott T. Aaronson, M.D, Director, Clinical Research Programs, Sheppard Pratt Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14947483
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): 25mg of Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Open-label

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 25 mg of psilocybin under supportive conditions to adult participants with BP-II, current episode depressed, in improving depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Bipolar Disorder (BP-II) Depression

Exclusion Criteria:

* Comorbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | From Baseline (Day -1) to three weeks post-dose.
  MADRS is a clinician-rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity. Response = >50% decrease and Remission =< 10 actual score

CONTACTS AND LOCATIONS:
Overall Officials: Scott Aaronson, MD, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No